CLINICAL TRIAL: NCT06055348
Title: A Phase Ib/II Clinical Study on the Safety, Pharmacokinetic Characteristics, and Preliminary Efficacy of SC0191 Combination Chemotherapy in Patients With Advanced Ovarian Cancer.
Brief Title: SC0191 Plus Chemotherapy in Advanced Ovarian Canceradvanced Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC0191-102
Record Dates: First submitted 2023-08-15; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Serous Ovarian Cancer; Advanced Ovarian Cancer
MeSH Terms: interventions — Drug Evaluation; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (SC0191 + Gemcitabine). (Experimental): SC0191 PO will be taken on days 1-3, 8-10, and 15-17 of each 28 day cycle. Gemcitabine 1000 mg/m² will be administered IV on days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: SC0191; Drug: Gemcitabine
- Arm B (SC0191 + Paclitaxel). (Experimental): SC0191 PO will be taken on days 1-3, 8-10, and 15-17 of each 28 day cycle. Paclitaxel 80 mg/m² will be administered IV on days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: SC0191; Drug: Paclitaxel

INTERVENTIONS:
Drug: SC0191 — SC0191 PO will be taken on days 1-3, 8-10, and 15-17 of each 28 day cycle.
  Other Names: Study drug
Drug: Gemcitabine — Gemcitabine 1000 mg/m² will be administered IV on days 1, 8, and 15 of each 28 day cycle.
  Other Names: Gemcitabine Injection
  Arms: Arm A (SC0191 + Gemcitabine).
Drug: Paclitaxel — Paclitaxel 80 mg/m² will be administered IV on days 1, 8, and 15 of each 28 day cycle.
  Other Names: Taxol
  Arms: Arm B (SC0191 + Paclitaxel).

SUMMARY:
A phase Ib/II clinical study on the safety, pharmacokinetic characteristics, and preliminary efficacy of SC0191 combination chemotherapy in patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
The phase 1b/2,multicenter, open-label study, contains 2 parts.

Part 1 Dose Escalation of SC0191 combination chemotherapy:

Part 1 will estimate the RP2D in dose escalation cohorts in patients withadvanced ovarian cancer.

Part 2 Dose Expansion of SC0191 plus Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced ovarian cancer that has failed or intolerant or not applicable to standard treatment (applicable to the dose escalation phase of stage Ib);
2. Histologically or cytologically confirmed advanced high-grade serous ovarian cancer, platinum-resistant or platinum-refractory recurrent ovarian cancer (applicable to the dose expansion phase of stage II);
3. There is at least one measurable lesion that meets the definition of RECIST 1.1;
4. Voluntarily participate in clinical trials and sign informed consent;
5. Age ≥18 years;
6. ECOG score of 0 to 1;
7. Predicted life expectancy ≥3 months;
8. Adequate bone marrow, liver biochemistry, renal function, and coagulation status.
9. Female patients who agree to use adequate contraceptive measures.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, immunotherapy or biological therapy, steroid therapy or other investigational drugs <28 days prior to the first dose of study treatment.
2. Patients who have not fully recovered from surgery according to the investigator's judgment.;
3. Patients who have previously received WEE1 inhibitor treatment;
4. Unresolved AEs or toxicities due to previous treatments;
5. Patients with contraindications or a history of severe allergies to gemcitabine or paclitaxel;
6. Known malignant CNS disease other than neurologically stable, treated brain metastases;
7. Other medical conditions or systemic diseases not suitable to participate;
8. The need for long-term therapeutic doses of anticoagulant or antiplatelet drugs;
9. Received CYP3A4 moderate or strong inhibitors or CYP3A4 moderate or strong inducers within 14 days;
10. Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of SC0191 in combination with gemcitabine or paclitaxel | From the first dose of study treatment until 30 days after the last dose.
  ncidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
To identify the recommended Phase 2 dose (RP2D) of SC0191 in combination with gemcitabine or paclitaxel | Through Cycle 1 (cycle is 28 days）
  Incidence and severity of dose-limiting toxicities (DLTs) in DLT-evaluable subjects during Cycle 1

SECONDARY OUTCOMES:
To investigate the plasma pharmacokinetics (PK) of SC0191 in combination with gemcitabine or paclitaxel | Through Cycle 1 (cycle is 28 days）
  Plasma pharmacokinetics (PK) of SC0191 in combination with chemotherapy: Single Dose SC0191 Cmax, Tmax, t1/2,AUC0-24h, AUC0-last, CL/F, Vd/F, and steady state SC0191 Ctrough, Cmax,ss, Cavg,ss, Tmax,ss, AUC0-τ, Rac.
To obtain estimates of clinical activity by determining the objective response rate (ORR) of SC0191 in combination with gemcitabine or paclitaxel | Through completion
  Objective response rate (ORR) as defined by Response Evaluation Criteria in Solid Tumors RECIST version 1.1
To obtain estimates of clinical activity by determining the time to CA125 progression of SC0191 in combination with gemcitabine or paclitaxel | Through completion
  Time to CA125 progression according to the Gynecologic Cancer Intergroup (GCIG) criteria
To obtain estimates of clinical activity by determining the progression-free survival (PFS) of SC0191 in combination with gemcitabine or paclitaxel | Through completion
  Progression-free survival (PFS) as defined by RECIST version 1.1 and clinical criteria
To obtain estimates of clinical activity by determining the duration of response (DOR) of SC0191 in combination with gemcitabine or paclitaxel | Through completion
  Duration of response (DOR) as defined by Response Evaluation Criteria in Solid Tumors RECIST version 1.1
To obtain estimates of clinical activity by determining the disease control rate (DCR) of SC0191 in combination with gemcitabine or paclitaxel | Through completion
  Disease control rate (DCR) as defined by Response Evaluation Criteria in Solid Tumors RECIST version 1.1